CLINICAL TRIAL: NCT04268771
Title: A Randomized, Double-blind, Parallel Group, Multicenter Study to Assess the Immunogenicity and Safety of Transitioning Subjects With Rheumatoid Arthritis to Biosimilar Rituximab (DRL_RI) or Continued Treatment With Rituxan® or MabThera®
Brief Title: A Phase III Transition Study of DRL Rituximab to Reference Medicinal Products
Acronym: RI-01-007
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Dr. Reddy's Laboratories Limited (Industry)
Collaborators: PPD Development, LP (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RI-01-007
Record Dates: First submitted 2020-01-31; First posted 2020-02-13 (Actual); Results first posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-10

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Intervention Model Description: A randomized, double-blind, parallel group, multicenter study to assess the immunogenicity and safety of transitioning subjects with rheumatoid arthritis to biosimilar rituximab (DRL_RI) or continued treatment with Rituxan® or MabThera®
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A: DRL_RI (Experimental): Subjects who have already received at least 1 full course comprising two 1000 mg infusions of either US-rituximab or EU-rituximab and are candidates for re-treatment with Rituximab, will be enrolled. DRL_RI will be administrated in combination with MTX as two 1000 mg infusions on Day 1 and Day 15
  Interventions: Biological: Experimental: Arm A: DRL_RI
- Arm B: US-Rituximab or EU-Rituximab (Active Comparator): Subjects who have already received at least 1 full course comprising two 1000 mg infusions of either US-rituximab or EU-rituximab and are candidates for re-treatment with rituximab, will be enrolled.
  Patients enrolled in Arm -B will continue to receive US-rituximab or EU-rituximab. The rituximab reference product used (US-licensed rituximab [Rituxan] or EU-approved rituximab [MabThera]) should be the same in the prior and the randomized treatment course, respectively.
  Interventions: Biological: Arm B: Rituxan®/Mabthera®

INTERVENTIONS:
Biological: Experimental: Arm A: DRL_RI — Proposed rituximab biosimilar, 100mg or 500mg, concentrate for solution for infusion
  Arms: Arm A: DRL_RI
Biological: Arm B: Rituxan®/Mabthera® — Reference product US- rituximab (Rituxan®) or EU-rituximab (MabThera®), 100mg or 500mg, concentrate for solution for infusion
  Arms: Arm B: US-Rituximab or EU-Rituximab

SUMMARY:
The objective of the current study is to assess the immunogenicity and safety of transitioning subjects with RA to DRL_RI from US-rituximab/EU-rituximab to continued treatment with US-rituximab/EU-rituximab.

The primary objective of this study is to assess the immunogenicity of transitioning subjects with RA to DRL_RI (biosimilar rituximab) from US-rituximab/EU-rituximab to continued treatment with US-rituximab/EU-rituximab

To assess the safety of transitioning subjects with RA to DRL_RI from US-rituximab/EU-rituximab to continued treatment with US-rituximab/EU-rituximab.

DETAILED DESCRIPTION:
This is a randomized, double-blind, parallel group, multicenter, Phase 3 transition study in subjects with active RA who are eligible for the subsequent treatment course with US-rituximab or EU-rituximab according to the clinical judgment of the investigator.

Subjects will then be randomized by interactive web response system (IWRS) to receive either two 1000 mg infusions of DRL_RI (Arm A) or US-rituximab/EU-rituximab (Arm B) on Day 1 and Day 15.

Subjects randomized to Arm A will receive DRL_RI and subjects randomized to Arm B will continue to receive either US-rituximab or EU-rituximab.

The study will consist of a screening period (Days -14 to 0) and a double-blind period (Day 1 to Week 12). Subjects will attend a screening visit followed by a visit at Weeks 0 (Day 1), 2, 4, 8, and 12 after randomization

It is planned that approximately 50 sites will be initiated for this study in up to 7 countries (including but not restricted to United States). There has been no randomization of patients till date for this study.

The study endpoints include:

The immunogenicity endpoint is:

• The incidence of anti-drug antibodies (ADA), including titer and neutralizing antibodies (NAb).

The primary safety endpoints are:

* Incidence of treatment-emergent adverse events (TEAEs) and serious adverse events (SAEs).
* Incidence of anaphylactic reactions, hypersensitivity reactions, and IRRs.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects aged 18 years or older who have provided valid written informed consent.
2. Subjects with a diagnosis of active RA who are eligible for the subsequent treatment course with US-rituximab or EU-rituximab according to the clinical judgment of the investigator.
3. Documented evidence that subject has received at least 1 full course comprising two 1000 mg infusions of either US-rituximab at least 16 weeks prior to the randomization visit or EU-rituximab at least 24 weeks prior to the day of randomization visit.
4. Subjects receiving a stable dose of weekly methotrexate (MTX) for at least 4 weeks prior to randomization (between 7.5 mg and 25 mg) and folic acid (at least 5 mg per week.

EXCLUSION CRITERIA;

1. Subjects with RA in functional Class IV
2. Subjects with human immunodeficiency virus (positive HIV1Ab or HIV2Ab), hepatitis B virus and/or hepatitis C virus infection, including those with positive results in the viral disease screening.
3. Subjects with active tuberculosis. Subjects with evidence of latent TB or a history of TB must have completed treatment or have initiated treatment for at least 1 month before the first dose of study treatment (Day 1). TB testing is required only if it is required by local regulations or practice.
4. Active systemic infection.
5. Severely immunocompromised.
6. History of severe hypersensitivity to either US-rituximab or EU-rituximab or any of its excipients requiring drug discontinuation.
7. Any serious illness or uncontrolled medical condition, including but not limited to severe infections, significant hepatic or renal disease, uncontrolled hypertension despite treatment (defined as blood pressure ≥160/95 mmHg), congestive heart failure (New York Heart Association [NYHA] Class III or IV), or other severe, uncontrolled cardiac disease or uncontrolled diabetes with immediate risk of acute complications.
8. Any condition that in the opinion of the investigator represents an obstacle for study conduct and/or represents a potential unacceptable risk for subjects.
9. Requires treatment with any biological medicinal product during the study other than the study treatment.
10. Previous treatment with B-cell modulating or cell depleting biologic therapy except US-rituximab or EU-rituximab.
11. Prior participation in this clinical trial or prior participation in any clinical trial with any monoclonal antibody within 12 months of screening or prior participation in any clinical trial within 3 months of screening or within 5 half-lives of the investigational drug or until the expected PD effect has returned to baseline, whichever is longer.
12. Treatment with other biologic disease-modifying anti-rheumatic drugs, or Janus kinase (JAK) inhibitors administered within 12 weeks before the first dose of rituximab of the prior treatment course onwards till the date of randomization.
13. Subjects with the following laboratory abnormalities:

    * Subjects with screening total white blood cell count <3000/μL, platelets <100,000/μL, neutrophils <1,500/μL, or hemoglobin <8.5 g/dL
    * Abnormal liver function tests such as aspartate aminotransferase, alanine aminotransferase, or alkaline phosphatase >2 × upper limit of normal (ULN). A single parameter >2 × ULN can be re-checked as soon as possible, at least prior to randomization, if required as per the investigator's discretion.
    * Creatinine clearance (Cockcroft & Gault formula) of less than 50 mL/min.
14. History of vaccination with live vaccines within 4 weeks of the first dose of study treatment (Day 1) or known to require live vaccines during the study.
15. Lactating or pregnant female.
16. Women of childbearing potential who do not consent to use highly effective methods of birth control (e.g., barrier contraceptives, oral contraceptives, intrauterine devices, true abstinence if it allowed as per the country specific regulatory requirement [periodic abstinence {e.g., calendar ovulation, symptothermal, post-ovulation methods} and withdrawal are not acceptable methods of contraception], or sterilization) during treatment and for at least 12 months after the last administration of study treatment.
17. For men involved in any sexual intercourse that could lead to pregnancy, subjects must agree to use 1 of the highly effective methods of birth control listed in Exclusion Criterion #16 during treatment and for at least 12 months after the last administration of study treatment.
18. Subject with serum IgG < lower limit of normal.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2020-04-08 (Actual); Primary Completion 2022-01-26 (Actual); Study Completion 2022-04-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (26):
- United States (26):
  - Arizona Arthritis and Rheumatology Research, PLLC, Phoenix, Arizona
  - California Allergy and Asthma Medical Group - CRN - PPDS 41230 11th Street West, Suite A, Palmdale, California
  - Inland Rheumatology Clinical Trials Incorporated, Upland, California
  - Rheumatology Consultant of Delaware dba Delaware Arthritis, Lewes, Delaware
  - MedBio Trials, Aventura, Florida
  - Clinical Research of West Florida Inc - Clearwater, Clearwater, Florida
  - Medical Research Center, Miami, Florida
  - AppleMed Research Group, LLC, Miami, Florida
  - Integral Rheumatology and Immunology Specialist, 140 Southwest 84th Avenue, Suite B, Plantation, Florida
  - Vicis Clinical Research INC, Tampa, Florida
  - Springfield Clinic (Clinic location), Springfield, Illinois
  - Bluegrass Community Research Inc,330 Waller Avenue, Suite 100,, Lexington, Kentucky
  - Arthritis and Osteoporosis Associates, Freehold, New Jersey
  - Integrative Rheumatology, Charlotte, North Carolina
  - Altoona Center For Clinical Research, 175 Meadowbrook Lane,, Duncansville, Pennsylvania
  - Articularis Healthcare Group, Inc dba Low Country Rheumatology, Summerville, South Carolina
  - Accurate Clinical Management, LLC, Baytown, Texas
  - Trinity Clinical Research LLC, 2008 East Hebron Parkway, Suites 120/114/100,, Carrollton, Texas
  - Abigail Neiman, Houston, Texas
  - Accurate Clinical Management, LLC, Houston, Texas
  - Laila A Hassan, MD, PA, Houston, Texas
  - Accurate Clinical Research-Houston, 11003 Resource Parkway, Suite 102, Houston, Texas
  - Houston Rheumatology & Arthritis Specialists, Katy, Texas
  - Clinical Associates in Research Therapeutics of America, LLC, San Antonio, Texas
  - Accurate Clinical Research, Inc., San Antonio, Texas
  - Accurate Clinical Research-League City, Texas City, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm B: US-Rituximab or EU-Rituximab: Subjects who have already received at least 1 full course comprising two 1000 mg infusions of either US-rituximab or EU-rituximab and are candidates for re-treatment with rituximab, will be enrolled.
  Patients enrolled in Arm -B will continue to receive US-rituximab or EU-rituximab. The rituximab reference product used (US-licensed rituximab [Rituxan] or EU-approved rituximab [MabThera]) should be the same in the prior and the randomized treatment course, respectively.
  Arm B: Rituxan®/Mabthera®: Reference product US- rituximab (Rituxan®) or EU-rituximab (MabThera®), 100mg or 500mg, concentrate for solution for infusion
Period: Overall Study
Arm/Group | Arm A: DRL_RI | Arm B: US-Rituximab or EU-Rituximab
Started | 70 | 70
Completed | 66 | 68
Not Completed | 4 | 2

BASELINE CHARACTERISTICS:
Population: Baseline analysis population include all the randomized study Participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: DRL_RI | Arm B: US-Rituximab or EU-Rituximab | Total
Number analyzed (Participants) | 70 | 70 | 140
Age, Categorical [Count of Participants; unit: Participants] — Population: Study Participants
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 47 | 39 | 86
    >=65 years | 23 | 31 | 54
Sex: Female, Male [Count of Participants; unit: Participants] — Study Participants
  Participants
    Female | 54 | 61 | 115
    Male | 16 | 09 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 5 | 12
  Not Hispanic or Latino | 60 | 64 | 124
  Unknown or Not Reported | 3 | 1 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 69 | 70 | 139
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants] — study participants regional distribution globally was reported here
  participants
    United States | 23 | 22 | 45
    Europe | 47 | 48 | 95
Time from prior rituximab [Mean (Standard Deviation); unit: months] — The time period in months for which duration the subjects had received the reference treatment (Rituxan or MabThera)
  months | 7.5 (2.65) | 7.6 (2.85) | 7.6 (2.77)

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Positive Anti-Drug Antibodies (ADA) on Day 1
Description: For Immunogenicity: Number of subjects with positive Anti-Drug Antibodies (ADA) on Day 1 was reported
Time Frame: ADA will be obtained before the administration of study treatment on Day 1
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: DRL_RI | Arm B: US-Rituximab or EU-Rituximab
Number analyzed (Participants) | 69 | 68
Participants | 3 | 1

2. Primary Outcome: Number of Subjects With Positive Anti-Drug Antibodies (ADA) on Day 15
Description: For Immunogenicity: Number of subjects with positive Anti-Drug Antibodies (ADA) on Day 15 was reported
Time Frame: ADA will be obtained before the administration of study treatment on Day 15
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: DRL_RI | Arm B: US-Rituximab or EU-Rituximab
Number analyzed (Participants) | 69 | 68
Participants | 1 | 0

3. Primary Outcome: Number of Subjects With Positive Anti-Drug Antibodies (ADA) at Week 4
Description: For Immunogenicity: Number of subjects with positive Anti-Drug Antibodies (ADA) at Week 4 was reported
Time Frame: ADA will be obtained before the administration of study treatment at Week 4
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: DRL_RI | Arm B: US-Rituximab or EU-Rituximab
Number analyzed (Participants) | 69 | 68
Participants | 0 | 0

4. Primary Outcome: Number of Subjects With Positive Anti-Drug Antibodies (ADA) at Week 8
Description: For Immunogenicity: Number of subjects with positive Anti-Drug Antibodies (ADA) at Week 8 was reported
Time Frame: ADA will be obtained before the administration of study treatment at Week 8
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: DRL_RI | Arm B: US-Rituximab or EU-Rituximab
Number analyzed (Participants) | 69 | 68
Participants | 1 | 0

5. Primary Outcome: Number of Subjects With Positive Anti-Drug Antibodies (ADA) at Week 12 Visits
Description: For Immunogenicity: Number of subjects with positive Anti-Drug Antibodies (ADA) at Week 12 visits was reported
Time Frame: ADA will be obtained at Week 12
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: DRL_RI | Arm B: US-Rituximab or EU-Rituximab
Number analyzed (Participants) | 69 | 68
Participants | 1 | 2

6. Secondary Outcome: Number of Subjects Reporting Anaphylactic Reactions at Dosing Time Points (Either at Week 1 or Week 3)
Description: Number of Subjects reporting anaphylactic reactions during the study drug administration either at Week 1 or Week 3 was reported
Time Frame: Assessments of Anaphylactic reactions will be carried out at either Week 1 or Week 3
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: DRL_RI | Arm B: US-Rituximab or EU-Rituximab
Number analyzed (Participants) | 70 | 70
Participants | 0 | 0

7. Secondary Outcome: Number of Subjects Reporting TEAEs (Treatment Emergent Adverse Events) That Led to Study Drug Discontinuation at Either Week 1 or Week 3 Dosing Timepoint
Description: TEAEs (Treatment emergent adverse events) which lead to study subjects discontinuation from the study drug administration at either week 1 or week 3 dosing timepoint
Time Frame: Assessment of AE's (Adverse Events) that led to study drug discontinuation were carried out at either week 1 or week 3 dosing timepoint
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: DRL_RI | Arm B: US-Rituximab or EU-Rituximab
Number analyzed (Participants) | 70 | 70
Participants | 1 | 1

8. Secondary Outcome: Number of Subjects Reporting SAEs (Serious Adverse Events) From Baseline (Week 1) to End of Study (Week 26)
Description: Incidence of SAEs: SAE is defined as "Results in death, is life-threatening, Requires in-subject hospitalization or prolongs existing hospitalization, Results in persistent or significant disability/incapacity".
  The measure here is only subjects reporting SAE.
Time Frame: Assessment of SAE's was carried out from baseline (week 1) to end of study (week 26)
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: DRL_RI | Arm B: US-Rituximab or EU-Rituximab
Number analyzed (Participants) | 70 | 70
Participants | 4 | 2

9. Secondary Outcome: Number of TEAEs Reported From Baseline (Week 1) to End of Study (Week 26)
Description: Number of TEAEs: Treatment-emergent AE are defined as any AE occurring or worsening on or after the first dose of study medication.
Time Frame: Assessment of AE's will be carried out from baseline (week 1) to end of study (week 26)
Population: Safety population
Measure: Number; unit: Number of events
Units Other Than Participants: Events
Arm/Group | Arm A: DRL_RI | Arm B: US-Rituximab or EU-Rituximab
Number analyzed (Participants) | 70 | 70
Number analyzed (Events) | 37 | 54
Number of events | 35 | 54

10. Secondary Outcome: Number of Subjects Reporting AE From Baseline (Week 1) to End of Study (Week 26)
Description: number of subjects reporting AE in the overall study are defined as any AE occurring or worsening after the ICF signed in the study
Time Frame: Assessment of AE's will be carried out from baseline (week 1) to end of study (week 26)
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: DRL_RI | Arm B: US-Rituximab or EU-Rituximab
Number analyzed (Participants) | 70 | 70
Participants | 24 | 27

11. Secondary Outcome: Number of Subjects Reporting TEAEs From Baseline (Week 1) to End of Study (Week 26)
Description: Number of subjects reporting Treatment-emergent AE (TEAEs) are defined as any AE occurring or worsening on or after the first dose of study medication.
Time Frame: Assessment of AE's will be carried out from baseline (week 1) to end of study (week 26)
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: DRL_RI | Arm B: US-Rituximab or EU-Rituximab
Number analyzed (Participants) | 70 | 70
Participants | 24 | 27

12. Secondary Outcome: Number of Subjects Reporting Hypersensitivity Reactions at Dosing Time Points (Either at Week 1 or Week 3)
Description: Safety assessment will be done by measuring hypersensitivity reactions at Dosing Time Points (Either at Week 1 or Week 3)
Time Frame: Assessments of hypersensitivity reactions either at Week 1 or Week 3
Measure: Number; unit: participants
Arm/Group | Arm A: DRL_RI | Arm B: US-Rituximab or EU-Rituximab
Number analyzed (Participants) | 70 | 70
participants | 0 | 1

13. Secondary Outcome: Number of Subjects Reporting Infusion-related Reactions (IRRs) at Dosing Time Points (Either at Week 1 or Week 3)
Description: Safety assessment: Number of Subjects Reporting Infusion-related reactions (IRRs) at Dosing Time Points (Either at Week 1 or Week 3) was reported
Time Frame: Assessments of IRRs were carried out at either Week 1 or Week 3
Population: Safety population
Measure: Number; unit: participants
Arm/Group | Arm A: DRL_RI | Arm B: US-Rituximab or EU-Rituximab
Number analyzed (Participants) | 70 | 70
participants | 2 | 0

ADVERSE EVENTS:
Time Frame: Till week 26
Arm/Group | Arm A: DRL_RI | Arm B: US-Rituximab or EU-Rituximab
All-Cause Mortality (participants affected / at risk) | 4/70 | 2/70
Serious Adverse Events (participants affected / at risk) | 4/70 | 2/70
Other Adverse Events (participants affected / at risk) | 3/70 | 17/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: DRL_RI (N=70) | Arm B: US-Rituximab or EU-Rituximab (N=70)
Myocardial Infarction (Cardiac disorders) | 1 (1) | 0 (0)
Intestinal resection (Surgical and medical procedures) | 1 (1) | 0 (0)
Embolic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
COVID-19 Pneumonia (Infections and infestations) | 2 (2) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 1 (1)
Empyema (Infections and infestations) | 0 (0) | 1 (1)
Septic Shock (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: DRL_RI (N=70) | Arm B: US-Rituximab or EU-Rituximab (N=70)
Headache (Nervous system disorders) | 0 (0) | 5 (5)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 5 (5)
COVID-19 (Infections and infestations) | 1 (1) | 4 (4)
Nasopharyngitis (Infections and infestations) | 0 (0) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2020-07-10): https://cdn.clinicaltrials.gov/large-docs/71/NCT04268771/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-16): https://cdn.clinicaltrials.gov/large-docs/71/NCT04268771/SAP_001.pdf